CLINICAL TRIAL: NCT04492189
Title: Impact of Containment Measures in People With Eating Disorders: a Descriptive Study
Brief Title: Containment Measures and Eating Disorders
Acronym: COVITA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: INSERM U1061 (Statistics) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0220
Record Dates: First submitted 2020-04-19; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-06

CONDITIONS: Eating Disorders; COVID 19
MeSH Terms: conditions — Feeding and Eating Disorders; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since March 17, 2020, the French government has implemented national containment measures due to the COVID-19 epidemic. Quarantine is an unpleasant experience : Separation from relatives, loss of liberty, concern about the infectious status, boredom, can negatively affect mental health, with the emergence of anxiety and depressive symptoms.

In addition, confinement can disrupt usual physical activity, a major destabilization criterion for patients suffering from eating disorders (ED). Finally, conditions of confinement can harm social support, yet identified as a protective and resilience factor in stress contexts. Thus, the current context of confinement and social distances could be source of an increase in eating behavior disorders symptoms in people suffering from ED.

DETAILED DESCRIPTION:
Investigators will recruit 40 patients with eating disorders. All patients were initially assessed in the daily hospital of the Endocrinology, Diabetes, Nutrition Department (Montpellier University Hospital) from January to march 2020.

All participants will performed a phone interview to assess eating disorder symptoms, caracteristicus of containment, 1 month after the beginning of the containment, and 1 month after the end of the containment.

ELIGIBILITY:
Inclusion criteria:

* Adult women
* Surferring from ED
* Assessed in the ED daily hospital (UH of Montpellier) from January to March 2020

Exclusion criteria:

* minors
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients are adult women with a diagnostic of ED
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Variation in eating disorders | 1 month
  the investigators aim to investigate the link between containment measures
Variation in eating disorders | 1 month
  the investigators aim to investigate the link between ED symptomatology with EDE-Q (eating disorder evaluation, caractéristiques du TCA)

SECONDARY OUTCOMES:
Vision of the bodily aspect | 1 month
  The investigators aim to investigate the link between containment measures
Vision of the bodily aspect | 1 month
  The investigators aim to investigate the link between body dissatisfaction
Variation in physical activity | 1 month
  the investigators aim to investigate the link between containment measures
Variation in physical activity | 1 month
  the investigators aim to investigate the link between physical activity
Identify the clinical factors modulating the psychological state during confinement | 1 month
  the investigators aim to investigate the link between containment measures
Identify the clinical factors modulating the psychological state during confinement | 1 month
  the investigators aim to investigate the link between emotional eating

CONTACTS AND LOCATIONS:
Overall Officials: Ariane SULTAN, PR, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC